CLINICAL TRIAL: NCT02871752
Title: Reducing the Effects of Active Surveillance Stress, Uncertainty and Rumination Thru Engagement in Mindfulness Education
Acronym: REASSUREME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Fox Chase Cancer Center (Other); University of Michigan (Other); Endeavor Health (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Victorson, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STU00105259; R01CA193331-01A1 (NIH)
Record Dates: First submitted 2016-08-05; First posted 2016-08-18 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; active surveillance; MBSR; couples; health promotion; quality of life; mindfulness
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Health Promotion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR (Mindfulness condition) (Experimental): MBSR (mindfulness-based stress reduction) is a group-based, 8-week program that was developed at the University of Massachusetts Stress Reduction Clinic under the direction of Jon Kabat-Zinn. MBSR is comprised of a structured, developmentally sequenced curriculum that uses a group format to experientially instruct participants in the practice of mindfulness meditation and mindful Hatha yoga. Each session includes different forms of meditation practice, such as cultivating awareness of thoughts, feelings and bodily sensations, and learning to incorporate this awareness during stressful emotional and/or physical life situations. Lesson activities include the following: (1) mindful meditation (e.g., awareness of breathing, body scan, sitting, walking); (2) yoga; and (3) group discussion.
  Interventions: Behavioral: Health promotion
- HealthPro (Control Matched Condition) (Active Comparator): HealthPro is a health promotion program designed by Dr. David Victorson of Northwestern University Medical Social Sciences Department and his research team to function as a matched control for the MBSR intervention in this research study. The program teaches and promotes healthy behaviors, skills, and lifestyles. Major learning themes include: (1) health behavioral change readiness and self-assessment; (2) physical activity, movement, and non-sedentary lifestyles; (3) dietary and nutritional considerations for optimal health; (4) emotional wellness and coping with difficulties; (5) social engagement, relationships intimacy, and health; (6) managing bodily pain; (7) weight management and weight loss strategies; (8) health behavior maintenance over the long-term.
  Interventions: Behavioral: Health promotion

INTERVENTIONS:
Behavioral: Health promotion — mindfulness-based stress reduction

SUMMARY:
We propose to examine the efficacy of couples-based mindfulness-based stress reduction (MBSR) on positive and negative psychological responses to active surveillance (AS) and AS adherence, with a sample of men on AS and their spouses.

DETAILED DESCRIPTION:
The current study proposes to examine the efficacy of couples-based mindfulness-based stress reduction (MBSR) on positive and negative psychological responses to active surveillance (AS) and AS adherence, with a larger, more geographically representative sample of men on AS and their spouses. We will compare the MBSR intervention condition (Group A) with a health promotion and wellness condition (Group B) in a sample of prostate cancer patients and their spouses. We will evaluate its efficacy on self-reported measures of positive and negative psychological responses to AS.

PRIMARY AIM Examine longitudinal change in positive and negative psychological responses to AS between groups over time.

SECONDARY AIM Observe the relation between positive and negative psychological responses to AS and AS adherence between groups over time.

THIRD AIM Explore dyadic factors on positive and negative psychological responses to AS and AS adherence between groups over time.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with prostate cancer and on active surveillance within the past 36 months (or the spouse or significant other of someone with prostate cancer on active surveillance)
* Must be at least 18 years of age
* Must be able to read, write, speak and understand English
* Must be able to perform basic activities of daily living (as determined by referring physician)
* Must be cognitively intact and free of serious psychiatric illness (as determined by referring physician)
* Must have access to the internet and ability to locate the assessment URL and/or ability to use a touchscreen keypad on a tablet device
* Must be willing to commit to the 8-week MBSR or Health Promotion course, which includes attending weekly, 2.5 hours classes over an 8 week period, a half-day retreat between week 6 and 7 , and daily homework assignments
* Must be willing to complete study assessments

Exclusion Criteria:

* Unable to provide consent
* Bedridden, or physical debilitation such that study participation would not be feasible or would create undue hardship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
longitudinal change in psychological responses as assessed through online survey | Baseline, Week 8, Month 6, Month 12
  longitudinal change in psychological responses as assessed through online survey

SECONDARY OUTCOMES:
relation between psychological responses to AS as assessed by online survey | Baseline, Week 8, Month 6, Month 12
  relation between psychological responses to AS as assessed by online survey
dyadic factors on psychological responses as assessed by online survey | Baseline, Week 8, Month 6, Month 12
  dyadic factors on psychological responses as assessed by online survey

CONTACTS AND LOCATIONS:
Overall Officials: David E Victorson, Ph.D., Principal Investigator — Northwestern University
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eton DT, Lepore SJ, Helgeson VS. Early quality of life in patients with localized prostate carcinoma: an examination of treatment-related, demographic, and psychosocial factors. Cancer. 2001 Sep 15;92(6):1451-9. doi: 10.1002/1097-0142(20010915)92:63.0.co;2-r. PMID 11745222
- [Background] Eton DT, Lepore SJ, Helgeson VS. Psychological distress in spouses of men treated for early-stage prostate carcinoma. Cancer. 2005 Jun 1;103(11):2412-8. doi: 10.1002/cncr.21092. PMID 15858824
- [Background] Eton DT, Lepore SJ. Prostate cancer and health-related quality of life: a review of the literature. Psychooncology. 2002 Jul-Aug;11(4):307-26. doi: 10.1002/pon.572. PMID 12203744
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Salminen EK, Portin RI, Koskinen AI, Helenius HY, Nurmi MJ. Estradiol and cognition during androgen deprivation in men with prostate carcinoma. Cancer. 2005 Apr 1;103(7):1381-7. doi: 10.1002/cncr.20962. PMID 15717315
- [Background] Krupski TL, Smith MR, Lee WC, Pashos CL, Brandman J, Wang Q, Botteman M, Litwin MS. Natural history of bone complications in men with prostate carcinoma initiating androgen deprivation therapy. Cancer. 2004 Aug 1;101(3):541-9. doi: 10.1002/cncr.20388. PMID 15274067
- [Background] Smith MR, McGovern FJ, Fallon MA, Schoenfeld D, Kantoff PW, Finkelstein JS. Low bone mineral density in hormone-naive men with prostate carcinoma. Cancer. 2001 Jun 15;91(12):2238-45. PMID 11413511
- [Background] Smith MR. Osteoporosis during androgen deprivation therapy for prostate cancer. Urology. 2002 Sep;60(3 Suppl 1):79-85; discussion 86. PMID 12231056
- [Background] Pirl WF, Siegel GI, Goode MJ, Smith MR. Depression in men receiving androgen deprivation therapy for prostate cancer: a pilot study. Psychooncology. 2002 Nov-Dec;11(6):518-23. doi: 10.1002/pon.592. PMID 12476433
- [Background] Dale W, Bilir P, Han M, Meltzer D. The role of anxiety in prostate carcinoma: a structured review of the literature. Cancer. 2005 Aug 1;104(3):467-78. doi: 10.1002/cncr.21198. PMID 15959911
- [Background] Cooperberg MR, Broering JM, Litwin MS, Lubeck DP, Mehta SS, Henning JM, Carroll PR; CaPSURE Investigators. The contemporary management of prostate cancer in the United States: lessons from the cancer of the prostate strategic urologic research endeavor (CapSURE), a national disease registry. J Urol. 2004 Apr;171(4):1393-401. doi: 10.1097/01.ju.0000107247.81471.06. PMID 15017184
- [Background] Roemeling S, Roobol MJ, Postma R, Gosselaar C, van der Kwast TH, Bangma CH, Schroder FH. Management and survival of screen-detected prostate cancer patients who might have been suitable for active surveillance. Eur Urol. 2006 Sep;50(3):475-82. doi: 10.1016/j.eururo.2006.04.019. Epub 2006 May 3. PMID 16713065
- [Background] Ganz PA, Barry JM, Burke W, Col NF, Corso PS, Dodson E, Hammond ME, Kogan BA, Lynch CF, Newcomer L, Seifter EJ, Tooze JA, Viswanath KV, Wessells H. NIH State-of-the-Science Conference Statement: Role of active surveillance in the management of men with localized prostate cancer. NIH Consens State Sci Statements. 2011 Dec 5-7;28(1):1-27. PMID 23392076
- [Background] Parker C. Active surveillance: towards a new paradigm in the management of early prostate cancer. Lancet Oncol. 2004 Feb;5(2):101-6. doi: 10.1016/S1470-2045(04)01384-1. PMID 14761814
- [Background] Parker C. Active surveillance of early prostate cancer: rationale, initial results and future developments. Prostate Cancer Prostatic Dis. 2004;7(3):184-7. doi: 10.1038/sj.pcan.4500720. PMID 15224088
- [Background] Bergman J, Litwin MS. Quality of life in men undergoing active surveillance for localized prostate cancer. J Natl Cancer Inst Monogr. 2012 Dec;2012(45):242-9. doi: 10.1093/jncimonographs/lgs026. PMID 23271780
- [Background] Kazer MW, Psutka SP, Latini DM, Bailey DE Jr. Psychosocial aspects of active surveillance. Curr Opin Urol. 2013 May;23(3):273-7. doi: 10.1097/MOU.0b013e32835eff24. PMID 23422588
- [Background] Carlson LE, Ursuliak Z, Goodey E, Angen M, Speca M. The effects of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients: 6-month follow-up. Support Care Cancer. 2001 Mar;9(2):112-23. doi: 10.1007/s005200000206. PMID 11305069
- [Background] Astin JA. Stress reduction through mindfulness meditation. Effects on psychological symptomatology, sense of control, and spiritual experiences. Psychother Psychosom. 1997;66(2):97-106. doi: 10.1159/000289116. PMID 9097338
- [Background] Wong SY. Effect of mindfulness-based stress reduction programme on pain and quality of life in chronic pain patients: a randomised controlled clinical trial. Hong Kong Med J. 2009 Oct;15 Suppl 6:13-4. No abstract available. PMID 19801710
- [Background] Chiesa A, Serretti A. Mindfulness-based stress reduction for stress management in healthy people: a review and meta-analysis. J Altern Complement Med. 2009 May;15(5):593-600. doi: 10.1089/acm.2008.0495. PMID 19432513
- [Background] Ledesma D, Kumano H. Mindfulness-based stress reduction and cancer: a meta-analysis. Psychooncology. 2009 Jun;18(6):571-9. doi: 10.1002/pon.1400. PMID 19023879
- [Background] Bohlmeijer E, Prenger R, Taal E, Cuijpers P. The effects of mindfulness-based stress reduction therapy on mental health of adults with a chronic medical disease: a meta-analysis. J Psychosom Res. 2010 Jun;68(6):539-44. doi: 10.1016/j.jpsychores.2009.10.005. Epub 2009 Dec 9. PMID 20488270
- [Background] Kabat-Zinn, J., Full Catastrophe Living: Using the Wisdom of your Mind to Face Stress, Pain and Illness. 1990, New York: Dell Publishing.
- [Background] Kabat-Zinn J, Massion AO, Kristeller J, Peterson LG, Fletcher KE, Pbert L, Lenderking WR, Santorelli SF. Effectiveness of a meditation-based stress reduction program in the treatment of anxiety disorders. Am J Psychiatry. 1992 Jul;149(7):936-43. doi: 10.1176/ajp.149.7.936. PMID 1609875
- [Background] Vollestad J, Sivertsen B, Nielsen GH. Mindfulness-based stress reduction for patients with anxiety disorders: evaluation in a randomized controlled trial. Behav Res Ther. 2011 Apr;49(4):281-8. doi: 10.1016/j.brat.2011.01.007. Epub 2011 Jan 27. PMID 21320700
- [Background] Gross CR, Kreitzer MJ, Thomas W, Reilly-Spong M, Cramer-Bornemann M, Nyman JA, Frazier P, Ibrahim HN. Mindfulness-based stress reduction for solid organ transplant recipients: a randomized controlled trial. Altern Ther Health Med. 2010 Sep-Oct;16(5):30-8. PMID 20882729
- [Background] Gross CR, Kreitzer MJ, Reilly-Spong M, Wall M, Winbush NY, Patterson R, Mahowald M, Cramer-Bornemann M. Mindfulness-based stress reduction versus pharmacotherapy for chronic primary insomnia: a randomized controlled clinical trial. Explore (NY). 2011 Mar-Apr;7(2):76-87. doi: 10.1016/j.explore.2010.12.003. PMID 21397868
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress, and immune parameters in breast and prostate cancer outpatients. Psychosom Med. 2003 Jul-Aug;65(4):571-81. doi: 10.1097/01.psy.0000074003.35911.41. PMID 12883107
- [Background] Carlson LE, Garland SN. Impact of mindfulness-based stress reduction (MBSR) on sleep, mood, stress and fatigue symptoms in cancer outpatients. Int J Behav Med. 2005;12(4):278-85. doi: 10.1207/s15327558ijbm1204_9. PMID 16262547
- [Background] Matousek RH, Dobkin PL, Pruessner J. Cortisol as a marker for improvement in mindfulness-based stress reduction. Complement Ther Clin Pract. 2010 Feb;16(1):13-9. doi: 10.1016/j.ctcp.2009.06.004. Epub 2009 Jul 4. PMID 20129404
- [Background] Matousek RH, Pruessner JC, Dobkin PL. Changes in the cortisol awakening response (CAR) following participation in mindfulness-based stress reduction in women who completed treatment for breast cancer. Complement Ther Clin Pract. 2011 May;17(2):65-70. doi: 10.1016/j.ctcp.2010.10.005. Epub 2010 Nov 26. PMID 21457893
- [Background] Carlson LE, Speca M, Patel KD, Goodey E. Mindfulness-based stress reduction in relation to quality of life, mood, symptoms of stress and levels of cortisol, dehydroepiandrosterone sulfate (DHEAS) and melatonin in breast and prostate cancer outpatients. Psychoneuroendocrinology. 2004 May;29(4):448-74. doi: 10.1016/s0306-4530(03)00054-4. PMID 14749092
- [Background] Lamanque P, Daneault S. [Does meditation improve the quality of life for patients living with cancer?]. Can Fam Physician. 2006 Apr;52(4):474-5. French. PMID 17327889
- [Background] Matchim Y, Armer JM. Measuring the psychological impact of mindfulness meditation on health among patients with cancer: a literature review. Oncol Nurs Forum. 2007 Sep;34(5):1059-66. doi: 10.1188/07.ONF.1059-1066. PMID 17878133
- [Background] Matchim Y, Armer JM, Stewart BR. Mindfulness-based stress reduction among breast cancer survivors: a literature review and discussion. Oncol Nurs Forum. 2011 Mar;38(2):E61-71. doi: 10.1188/11.ONF.E61-E71. PMID 21356643
- [Background] Ott MJ, Norris RL, Bauer-Wu SM. Mindfulness meditation for oncology patients: a discussion and critical review. Integr Cancer Ther. 2006 Jun;5(2):98-108. doi: 10.1177/1534735406288083. PMID 16685074
- [Background] Smith JE, Richardson J, Hoffman C, Pilkington K. Mindfulness-Based Stress Reduction as supportive therapy in cancer care: systematic review. J Adv Nurs. 2005 Nov;52(3):315-27. doi: 10.1111/j.1365-2648.2005.03592.x. PMID 16194185
- [Background] Saxe GA, Hebert JR, Carmody JF, Kabat-Zinn J, Rosenzweig PH, Jarzobski D, Reed GW, Blute RD. Can diet in conjunction with stress reduction affect the rate of increase in prostate specific antigen after biochemical recurrence of prostate cancer? J Urol. 2001 Dec;166(6):2202-7. PMID 11696736
- [Background] Pickles T, Ruether JD, Weir L, Carlson L, Jakulj F; SCRN Communication Team. Psychosocial barriers to active surveillance for the management of early prostate cancer and a strategy for increased acceptance. BJU Int. 2007 Sep;100(3):544-51. doi: 10.1111/j.1464-410X.2007.06981.x. Epub 2007 May 26. PMID 17532857
- [Result] Victorson D, Morgan T, Kutikov A, Novakovic K, Kundu S, Horowitz B, Jackson K, Addington E, Murphy K, Sauer C, Brendler C. Mindfulness-based stress reduction for men on active surveillance for prostate cancer and their spouses: Design and methodology of a randomized controlled trial. Contemp Clin Trials. 2023 Feb;125:107059. doi: 10.1016/j.cct.2022.107059. Epub 2022 Dec 21. PMID 36563902
- [Result] Schuette SAP, Cordero E, Slosburg K, Addington EL, Victorson D. A Scoping Review of Positive Lifestyle and Wellness Interventions to Inform the Development of a Comprehensive Health Promotion Program: "HealthPro". Am J Lifestyle Med. 2017 May 5;13(4):336-346. doi: 10.1177/1559827617704825. eCollection 2019 Jul-Aug. PMID 31285713